CLINICAL TRIAL: NCT03386916
Title: CT Scan Guide Percutaneous Biopsy of Lytic Bone Metastases of Lung Cancer : Pathology Diagnosis and Molecular Biology
Brief Title: CT Scan Guide Percutaneous Biopsy of Lytic Bone Metastases of Lung Cancer : Contribution in Pathology Diagnosis and Molecular Biology
Acronym: stasfa
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.218
Record Dates: First submitted 2017-12-12; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Image-Guided Biopsy - Carcinoma, Bronchogenic / Diagnosis- Outpatients
Keywords: Technology, Radiologic - Radiography, Interventional - Image-Guided Biopsy - Early Detection of Cancer - Carcinoma, Bronchogenic / diagnosis - Outpatients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with a CT scan guide percutaneous biopsy of lytic bone: Patient with a CT scan guide percutaneous biopsy of lytic bone metastases register on CHU Grenoble Alpes radiology software between January 2010 and June 2017
  Interventions: Procedure: CT scan guide percutaneous biopsy of lytic bone metastases of lung cancer

INTERVENTIONS:
Procedure: CT scan guide percutaneous biopsy of lytic bone metastases of lung cancer

SUMMARY:
In case of primary lung cancer, bone metastases biopsy can be done in initial diagnosis or follow-up.

Nevertheless, any study focus on rentability and biopsy complications of lytic bone lesion for the context of lung cancer.

This study aims to demonstrate that CT scan guide percutaneous biopsy of lytic bone lesion help to anatomopathologic diagnosis and molecular biology with a low complication rate inasmuch a lung cancer is suspected.

This study is observational, retrospective, one center

DETAILED DESCRIPTION:
Current progress in thoracic oncology require to be able to carry out analysis by molecular biology. So biopsies are done several times during cancer progression. But risk is high for a lung biopsy with enough sample, so a CT scan guide percutaneous biopsy of lytic bone metastases of lung cancer can be an alternative.

In case of primary lung cancer, bone metastases biopsy can be done in initial diagnosis or follow-up. But this contribution in diagnostic (anatomopathologic an molecular biology) is poorly understood. It is demonstrated that to sample on lytic bone lesion have a failure rate lower than on calcified osseous lesion. Nevertheless, any study focus on rentability and biopsy complications of lytic bone lesion for the context of lung cancer.

this study aims to demonstrate that CT scan guide percutaneous biopsy of lytic bone lesion help to anatomopathologic diagnosis and molecular biology with a low complication rate inasmuch a lung cancer is suspected.

This study is observational, retrospective, descriptive, one-center Patient's records selection will be done by keyword search on the CHU Grenoble Alpes radiology software. Only records with bone biopsy register between January 2010 and June 2017 will be included.

ELIGIBILITY:
Inclusion Criteria:

* CT scan guide percutaneous biopsy of lytic bone metastases
* register on CHU Grenoble Alpes radiology software between January 2010 and June 2017
* Patient who have a clinical context of lung cancer with bone metastases

Exclusion Criteria:

* Person deprived of liberty by judicial order
* Opposition expressed by patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CT scan guide percutaneous biopsy of lytic bone metastases of lung cancer
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Rentability of biopsy of lytic bone lesion in anatomopathologic analysis | Analysis between january 2018-september 2018
  Rentability of biopsy of lytic bone lesion = 100x (number of sample wich analysed by anatomopathologic /total number of biopsy of lytic bone lesion done)

SECONDARY OUTCOMES:
Rentability of biopsy of lytic bone lesion in molecular biology analysis inas much non small cell epidermoid lung cancer is diagnosed | Analysis between january 2018-september 2018
  Rentability of biopsy of lytic bone lesion in molecular biology analysis inas much non small cell epidermoid lung cancer is diagnosed
  - =100x (number of sample wich analysed by molecular biology /total number of biopsy of lytic bone lesion sent to molecular biology analysis)
Cell quality in sample of biopsy of lytic bone lesion in molecular biology analysis inas much non small cell epidermoid lung cancer is diagnosed | Analysis between january 2018-september 2018
  Cell quality in sample of biopsy of lytic bone lesion in molecular biology analysis inas much non small cell epidermoid lung cancer is diagnosed
  * average percentage of tumour cells in samples
Complication rate linked to gesture of biopsy of lytic bone lesion | Analysis between january 2018-september 2018
  Complication rate linked to gesture of biopsy of lytic bone lesion and descriptive analysis
Impact assessement of biopsy of lytic bone lesion on patient care | Analysis between january 2018-september 2018
  Modification of management of lung cancer between before biopsy and after biopsy results

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert FERRETTI, Study Director — UniversityHospital Grenoble

REFERENCES:
- [Background] Jelinek JS, Murphey MD, Welker JA, Henshaw RM, Kransdorf MJ, Shmookler BM, Malawer MM. Diagnosis of primary bone tumors with image-guided percutaneous biopsy: experience with 110 tumors. Radiology. 2002 Jun;223(3):731-7. doi: 10.1148/radiol.2233011050. PMID 12034942
- [Background] Fraser-Hill MA, Renfrew DL. Percutaneous needle biopsy of musculoskeletal lesions. 1. Effective accuracy and diagnostic utility. AJR Am J Roentgenol. 1992 Apr;158(4):809-12. doi: 10.2214/ajr.158.4.1546597.
- [Background] Leffler SG, Chew FS. CT-guided percutaneous biopsy of sclerotic bone lesions: diagnostic yield and accuracy. AJR Am J Roentgenol. 1999 May;172(5):1389-92. doi: 10.2214/ajr.172.5.10227522.
- [Background] Vieillard MH, Boutry N, Chastanet P, Duquesnoy B, Cotten A, Cortet B. Contribution of percutaneous biopsy to the definite diagnosis in patients with suspected bone tumor. Joint Bone Spine. 2005 Jan;72(1):53-60. doi: 10.1016/j.jbspin.2004.03.008. PMID 15681249
- [Background] Vanderlaan PA, Yamaguchi N, Folch E, Boucher DH, Kent MS, Gangadharan SP, Majid A, Goldstein MA, Huberman MS, Kocher ON, Costa DB. Success and failure rates of tumor genotyping techniques in routine pathological samples with non-small-cell lung cancer. Lung Cancer. 2014 Apr;84(1):39-44. doi: 10.1016/j.lungcan.2014.01.013. Epub 2014 Jan 28. PMID 24513263